CLINICAL TRIAL: NCT00141427
Title: Pregabalin In Partial Seizures (Preps) : An Open-Label, International, Multicenter Add-On Therapy Trial
Brief Title: Pregabalin In Partial Seizures: An Open-Label, International, Multicenter Add-On Therapy Trial.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081005
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2006-06

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To assess the clinical improvement (change in seizure frequency), safety and tolerability of patients with partial seizures following adjunctive therapy of pregabalin BID in addition to existing standard AEDs.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with a diagnosis of partial epilepsy.
* 18 years and older.

Exclusion Criteria:

* Having a treatable cause of seizure.
* Having a progressive neurological or systemic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540
Dates: Start 2004-11; Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Reduction in seizure frequency.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- Belgium (8):
  - Pfizer Investigational Site, Bruges
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Duffel
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Leuven
  - Pfizer Investigational Site, Liège
  - Pfizer Investigational Site, Tielt
  - Pfizer Investigational Site, Yvoir
- Finland (3):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kuopio
  - Pfizer Investigational Site, Tampere
- France (15):
  - Pfizer Investigational Site, Marseille, Cedex 05
  - Pfizer Investigational Site, Montpellier, Cedex 5
  - Pfizer Investigational Site, Lyon, Cedex
  - Pfizer Investigational Site, Bayonne
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Tours
- Netherlands (7):
  - Pfizer Investigational Site, The Hague, South Holland
  - Pfizer Investigational Site, Alkmaar
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Heeze
  - Pfizer Investigational Site, Hilversum
  - Pfizer Investigational Site, Oss
  - Pfizer Investigational Site, Southwest Heemstede
- Poland (5):
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Wroclaw
- Portugal (6):
  - Pfizer Investigational Site, Braga
  - Pfizer Investigational Site, Funchal
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Matosinhos Municipality
  - Pfizer Investigational Site, Ponta Delgada
  - Pfizer Investigational Site, Porto
- Switzerland (2):
  - Pfizer Investigational Site, Lausanne
  - Pfizer Investigational Site, Zurich
- United Kingdom (5):
  - Pfizer Investigational Site, Cambridge, Cambs
  - Pfizer Investigational Site, Truro, Cornwall
  - Pfizer Investigational Site, Plymouth, Devon
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Oxford
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081005&StudyName=Pregabalin+In+Partial+Seizures%3A+An+Open%2DLabel%2C+International%2C+Multicenter+Add%2DOn+Therapy+Trial%2E